CLINICAL TRIAL: NCT00640627
Title: A Double-Blind, Placebo-Controlled Study of the Efficacy and Tolerability of Once Daily Celebrex® (Celecoxib) vs. Placebo in the Treatment of Subjects With Osteoarthritis of the Knee Non-Responsive to Naproxen and Ibuprofen
Brief Title: Efficacy and Safety of Celecoxib Versus Placebo in the Treatment of Patients With Osteoarthritis of the Knee Who Were Unresponsive to Naproxen and Ibuprofen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191069
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsule once daily for 6 weeks
  Arms: A
Drug: Placebo — Matched oral placebo for 6 weeks
  Arms: B

SUMMARY:
To compare the safety and efficacy of celecoxib versus placebo in the treatment of patients with knee osteoarthritis who were unresponsive to treatment with prescription strength naproxen and ibuprofen or who could not tolerate prescription strength naproxen and ibuprofen

ELIGIBILITY:
Inclusion criteria:

* OA of the knee in flare state at baseline visit and functional capacity class of I-III
* Failed adequate trials of both naproxen and ibuprofen (prescription strength) within the past 5 years due to lack of efficacy, tolerability or both; duration of prescription strength ibuprofen and naproxen must have been a minimum of 2 weeks for each drug at the respective recommended doses if failure was due to lack of efficacy, and for any duration if failure was due to lack of tolerability

Exclusion criteria:

* Inflammatory arthritis or gout/pseudo-gout with acute flare within the past 2 years (subjects with fibrositis or fibromyalgia will not be excluded)
* Received acetaminophen within 24 hours of baseline visit
* Use of mobility assisting device for less than six weeks prior to study screening or use of a walker
* History of gastrointestinal (GI) perforation, obstruction, or bleeding
* Diagnosed or treated for GI ulcer within 60 days prior to first dose of study medication
* Recieved corticosteroids or hyaluronic acid within certain timeframe before study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2003-12; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Patient's Assessment of Arthritis Pain, according to visual analog scale (VAS) | Week 6

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | Week 6
Patient's and Physician's Global Assessment of Pain | Weeks 2 and 6
The Medical Outcomes Study Sleep Scale | Week 6
Adverse events | Weeks 0-6
Laboratory tests | Week 6
Vital signs | Week 6
Physical examination | Week 6
Patient's Assessment of Arthritis Pain according to VAS | Week 2
Serious adverse events | Up to 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Paramount, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Wheat Ridge, Colorado
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Woodstock, Georgia
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Chesterfield, Missouri
  - Pfizer Investigational Site, Reno, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Mason, Ohio
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Camp Hill, Pennsylvania
  - Pfizer Investigational Site, Jenkintown, Pennsylvania
  - Pfizer Investigational Site, Greensboro, South Carolina
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Murfreesboro, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Seattle, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191069&StudyName=A%20Double-Blind%2C%20Placebo-Controlled%20Study%20of%20the%20Efficacy%20and%20Tolerability%20of%20Once%20Daily%20Celebrex%C2%AE%20%28Celecoxib%29%20vs.%20Placebo%20in%20the%20Treatment%20of%20Subjects%20With%20Osteoarthritis%20of%20the%20Knee%20Non-Responsive%20to%20Naproxen%20and%20Ibuprofen